CLINICAL TRIAL: NCT06477029
Title: Modulating Ventral Striatal Activity and Connectivity With Transcranial Focused Ultrasound as a Putative Novel Intervention for Cocaine Use Disorder
Brief Title: Examination of Transcranial Focused Ultrasound on Brain Activity in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Phillips, MD MD (Cantab) (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Mary Phillips, MD MD (Cantab), Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY24020142; UG3DA060431 (NIH)
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Impulsive Behavior
Keywords: transcranial focused ultrasound; Magnetic Resonance Imaging; Reward
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VS tFUS/Sham tFUS (Experimental): VS tFUS (tFUS applied to the ventral striatum) Sham tFUS (go through the motions of applying tFUS to the VS)
  Interventions: Device: tFUS; Device: Sham tFUS
- Sham tFUS/VS tFUS (Experimental): VS tFUS (tFUS applied to the ventral striatum) Sham tFUS (go through the motions of applying tFUS to the VS)
  Interventions: Device: tFUS; Device: Sham tFUS

INTERVENTIONS:
Device: tFUS — tFUS is a brief stimulation of a part of the brain called the ventral striatum with low-intensity sound waves that pass through the scalp and skull safely.
Device: Sham tFUS — Sham tFUS goes through the motions of applying tFUS to the brain. Participants will know that one session will be a sham, but they will be blinded to which session is the sham

SUMMARY:
The investigators aim to examine the immediate effect of transcranial focused ultrasound (tFUS) on brain activity in healthy adults.

DETAILED DESCRIPTION:
The investigators will examine ventral striatum (VS) target engagement by tFUS in healthy adults using a reward processing task that reliably activates the VS.

ELIGIBILITY:
Inclusion Criteria:

* No present/lifetime history of major depressive disorder (MDD), psychosis, Bipolar Disorder; Hamilton Depression Rating Scale (HDRS)>7; Young Mania Rating Scale (YMRS)>10), borderline personality disorder, and present suicidal ideation
* No family history of MDD, psychosis, Bipolar Disorder, or epilepsy

Exclusion Criteria:

* Present/lifetime history of MDD, psychosis, Bipolar Disorder (HDRS>7; YMRS>10), borderline personality disorder, and present suicidal ideation. Childhood history of, but not present, anxiety disorders and Attention-deficit/hyperactivity disorder (ADHD) will be allowed as these are common disorders in childhood
* Family history of MDD, psychosis, Bipolar Disorder, or epilepsy
* History of head injury, neurological (e.g., epilepsy), pervasive developmental disorder (e.g., autism), systemic medical disease and treatment (medical records, participant report)
* Use of substances with seizure risk (e.g., stimulants) in the past month, as for other non-invasive neuromodulation techniques, assessed as screening and before each tFUS session
* Mini-Mental State Examination (MMSE) score (cognitive state) <24
* Premorbid North American Adult Reading Test (NAART) intelligence quotient (IQ) estimate <85;
* Visual disturbance: <20/40 (Snellen visual acuity)
* Left/mixed handedness (Annett criteria)
* History of alcohol or other substance use disorder (SUD), daily nicotine use, and/or illicit substance use over the last 3 months (SCID-5). Note: lifetime/present cannabis use (<3 times in the past month) at non-SUD levels will be allowed, given its common usage in young adults. Urine tests on scan days will exclude current illicit substance use. Salivary alcohol tests on scan days will exclude intoxicated individuals
* Binge drinking (as defined by National Institute on Alcohol Abuse and Alcoholism (NIAA) criteria: consuming 5 or more drinks (male), or 4 or more drinks (female), in about 2 hours.) in the week before, and/or >3 drinks/day for the 3 days before, and/or alcohol in the last 12 hrs before, any alcohol on tFUS scan day, confirmed at screening and scan days. Alcohol/nicotine/caffeine/cannabis use (below SCID-5 SUD and binge levels) will be allowed
* MRI exclusion criteria: metallic objects, e.g., surgical implants; claustrophobia; positive pregnancy test for females or self-report pregnancy
* Unable to understand English
* Taking any psychotropic medications in the past 3 months
* Any implanted neural device
* Color blind

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Ventral striatum (VS) activity to prediction error before receiving tFUS to the VS | Two visits over up to 8 weeks
  Measure of ventral striatum (VS) activity to prediction error before receiving tFUS to the VS
Ventral striatum (VS) activity to prediction error after receiving tFUS to the VS | Two visits over up to 8 weeks
  Measure of ventral striatum (VS) activity to prediction error after receiving tFUS to the VS

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Phillips, MD MD (Cantab), Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be available for access by the research community via National Institute of Mental Health Data Archive (NDA).
Time Frame: After each submission cycle, NDA conducts quality assurance (QA) procedures on submitted data during which access to data and images for research is temporarily suspended, typically a period lasting 4 months prior to sharing. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid findability. We will include DOI in relevant publications. NDA will decide how long to preserve the data, but has not deleted any deposited data to date.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.